CLINICAL TRIAL: NCT00392158
Title: Target-controlled Infusion of Propofol and Remifentanil During General Anaesthesia Guided by the Index Bispectral: Comparison Between Manual Perfusion and Automated Perfusion
Brief Title: Manual Administration of Propofol-remifentanil Versus Dual Closed-loop Using Bispectral Index as the Control Variable
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Foch-3
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Closed-loop anesthesia system

SUMMARY:
To compare manual administration of propofol and remifentanil and dual closed-loop using bispectral index as the control variable during anesthesia

DETAILED DESCRIPTION:
The Bispectral Index (BIS) is an electroencephalogram-derived measure of anesthetic depth. A closed-loop anesthesia system can be built using BIS as the control variable, a proportional-integral-differential control algorithm, and a propofol target-controlled infusion system as the control actuator. Recent studies have shown that such system is able to provide clinically adequate anesthesia. We hypothesized that BIS can also indicate the adequacy of analgesia and therefore built a combined closed-loop anesthesia system using BIS as the control variable, two proportional-integral-differential control algorithms, a propofol and a remifentanil target-controlled infusion systems as the control actuators. In preparation for a large multi-center control trial, we propose a prospective randomized study to evaluate the effectiveness of such a closed-loop anesthesia system. Two groups of patients are compared: one in which propofol and remifentanil are administered by the anesthesiologist using target-controlled infusion systems, and one in which propofol and remifentanil are administered automatically by the combined closed-loop anesthesia system. In both groups, the goal is to maintain BIS between 40 and 60, the recommended range during anesthesia by the manufacturer. We expect the combined closed-loop anesthesia system group to do similar or better.

ELIGIBILITY:
Inclusion Criteria:

* surgery under general anesthesia using relaxant agent,
* surgery lasting more than one hour

Exclusion Criteria:

* pregnant women,
* indication for rapid sequence induction,
* anticipation of difficult intubation,
* allergy to propofol or remifentanil,
* neurological or muscular disorder,
* combination of general anesthesia and of regional anesthesia,
* emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Global score (calculated parameter which depicts the performance of the system, i.e. its capacity to maintain BIS in the desired range)

SECONDARY OUTCOMES:
consumption of propofol and remifentanil during the induction and the maintenance of the anaesthesia
number of modifications of target of propofol and remifentanil
number of episodes of hemodynamic anomalies having required a treatment
intraoperative volume loading and transfusion
extubation time, explicit memorisation
dysfunctions of each system

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Principal Investigator — Hôpital Foch
Locations (6):
- France (6):
  - Dept of Anesthesia, CH d'Argenteuil, Argenteuil
  - Dept of Anesthesiology, CHU de Besançon, Besançon
  - Dept of Anesthesia, Clinique Saint Augustin, Bordeaux
  - Dept of Anesthesia and Intensive Care, Hôpital Beaujon, Clichy
  - Dept of Anesthesiology, Hôpital Cochin, Paris
  - Dept of Anesthesia, Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Background] Liu N, Chazot T, Trillat B, Pirracchio R, Law-Koune JD, Barvais L, Fischler M. Feasibility of closed-loop titration of propofol guided by the Bispectral Index for general anaesthesia induction: a prospective randomized study. Eur J Anaesthesiol. 2006 Jun;23(6):465-9. doi: 10.1017/S0265021506000196. PMID 16672092